CLINICAL TRIAL: NCT02855632
Title: The Efficacy of G-CSF Against Adhesion Reformation After Hysteroscopic Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Wenzhou people's hospital，zhejiang province,China (Unknown); Ningbo Women & Children's Hospital (Other)
Responsible Party: Principal Investigator, Xiaona Lin, MD, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SRRSHRMC2016001
Record Dates: First submitted 2016-04-03; First posted 2016-08-04 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Intrauterine Adhesion
Keywords: G-CSF; adhesion reformation; Asherman syndrome
MeSH Terms: conditions — Gynatresia | interventions — Granulocyte Colony-Stimulating Factor; Saline Solution; Sodium Chloride; Estrogens

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental): G-CSF(1.8ml) will be injected into the uterine cavity by insemination catheter 7 days after first hysteroscopic adhesiolysis.
  Interventions: Drug: G-CSF; Drug: hormone therapy; Other: Cook balloon
- Normal saline (Placebo Comparator): equal volume of normal saline(1.8ml) will be injected into the uterine cavity by insemination catheter 7 days after first hysteroscopic adhesiolysis.
  Interventions: Drug: Normal saline; Drug: hormone therapy; Other: Cook balloon

INTERVENTIONS:
Drug: G-CSF — 7 days after first hysteroscopic adhesiolysis, G-CSF will be injected into the uterine cavity after balloon removing.
  Other Names: granulocyte colony-stimulating factor
  Arms: G-CSF
Drug: Normal saline — 7 days after first hysteroscopic adhesiolysis, normal saline will be injected into the uterine cavity after balloon removing.
  Other Names: 0.9% NaCl; 0.9% sodium chloride
  Arms: Normal saline
Drug: hormone therapy — In all cases hormone therapy was commenced shortly after the operation, consisting of oestradiol valerate at a dose of 6 mg per day for 21-28 days with the addition of medroxyprogesterone acetate at a dose of 6 mg per day for the last 7-10 days of the oestrogen therapy. Following the withdrawal bleed, the hormone therapy was repeated for another cycle.
  Other Names: Artificial cycle; Artificial menstrual cycle; Estrogen and Progesterone Sequential Therapy
Other: Cook balloon — At the end of the procedure, the Cook balloon were placed in the uterine cavity of each patient.the device was removed after 7 days.

SUMMARY:
The purpose of this study is to investigate the efficacy of Granulocyte Colony Stimulating Factor(G-CSF) on decreasing adhesion reformation and improving fertility outcomes after hysteroscopic adhesiolysis in patients with moderate to severe intrauterine adhesions.

DETAILED DESCRIPTION:
After hysteroscopic adhesiolysis, patients with moderate to severe intrauterine adhesions will be allocated into 2 groups randomly, with COOK ballon and estrogen and progesterone sequential therapy given to prevent adhesion routinely. 7 day later, G-CSF or normal saline will be injected into the uterine cavity by Tom catheter after removing the balloon respectively. A second hysteroscopic examination will be performed in 2 months to check up the adhesion reformation. In addition, the endometrial thickness after surgery and fertility outcome will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and severe intrauterine adhesion patients(AFS score ≥5)
* age 18-40
* first time receiving hysteroscopic adhesiolysis
* provided COOK balloon as adjuvant adhesion prevention treatment
* accepting randomized trial

Exclusion Criteria:

* Mild adhesion patients
* uterine shape can't be restored in the end of surgery
* abnormal chromosome phenotype
* systemic disease
* no fertility desire
* contradiction of G-CSF injection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adhesion reformation rate | 2 months after first surgery
  Adhesion reformation rate after first adhesiolysis

SECONDARY OUTCOMES:
Pregnancy rate | 3 years after first surgery
  pregnancy rate after adhesiolysis
Live birth rate | 4 years after first surgery
  live birth rate after adhesiolysis

OTHER OUTCOMES:
Endometrial thickness | 1 months after G-CSF injection
  Endometrial thickness in the ovulation phase after G-CSF injection

CONTACTS AND LOCATIONS:
Overall Officials: Xiaona Lin, Doctor, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Chen X, Chen S, Wei C, Li B, Wang Z, Shen X, Lin X. Intrauterine administration of G-CSF for promoting endometrial growth after hysteroscopic adhesiolysis: a randomized controlled trial. Hum Reprod. 2022 Apr 1;37(4):725-733. doi: 10.1093/humrep/deac023. PMID 35147195